CLINICAL TRIAL: NCT06191679
Title: Decision Aid for Education and Support About Cancer Treatment
Acronym: DECIDES B+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-017521
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Childhood Cancer
Keywords: AYA
MeSH Terms: conditions — Neoplasms | interventions — Decision Support Techniques; Educational Status

STUDY DESIGN:
Intervention Model Description: Family Units (AYA and caregiver participants) are randomized to one of three arms:
  1. No intervention (referred to as "Usual Care")
  2. DECIDES with an informational handout (referred to as "DECIDES")
  3. DECIDES with coach-assisted support (referred to as "DECIDES+")
  Oncology Clinicians of participating AYA are not randomized to an intervention arm; they are enrolled to complete a singular Qualitative Interview to provide feedback for future implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Subjects will not receive the intervention and will only receive standard of care (i.e., subjects will access their health care team for decision support, per usual).
- DECIDES with Informational Handout (DECIDES) (Experimental): Subjects will receive access to the decision support intervention (DECIDES) along with an informational handout that includes goals of the decision support intervention and instructions for accessing the web-based application independently.
  Interventions: Behavioral: Decision Aid for Education and Support about Cancer Treatment (DECIDES Intervention)
- DECIDES with Coach-Assisted Support (DECIDES+) (Experimental): Subjects will receive access to the decision support intervention (DECIDES) along with live coach-assisted support for accessing and navigating the web-based application.
  Interventions: Behavioral: Decision Aid for Education and Support about Cancer Treatment (DECIDES Intervention)

INTERVENTIONS:
Behavioral: Decision Aid for Education and Support about Cancer Treatment (DECIDES Intervention) — DECIDES is a developmentally appropriate, engaging, and interactive web-based decision support intervention for AYA diagnosed with cancer (and their caregivers) that includes components written for low health literacy. Components include:
  * Education on cancer and cancer treatments, including clinical trials
  * An exercise to identify perceived barriers and benefits to treatment options
  * An exercise to clarify personal goals for treatment that align with life goals
  * Resources to support communication with the oncology health care team
  Arms: DECIDES with Coach-Assisted Support (DECIDES+); DECIDES with Informational Handout (DECIDES)

SUMMARY:
The goals of this clinical trial are to evaluate DECIDES, a web-based decision support application that provides education about cancer and cancer treatment and provides support to encourage adolescent and young adult (AYA) patients, their caregivers, and oncology health care providers to make informed decisions about cancer treatment together.

The main questions this study aims to answer are:

* Is DECIDES acceptable, usable, and feasible for AYA, caregivers, and oncology health care providers?
* Is DECIDES helpful for AYA, caregivers, and oncology health care providers that are making cancer treatment decisions together?

AYA and caregiver participants will complete a questionnaire and be randomly assigned to participate in one of three groups: (1) Usual Care, (2) DECIDES, or (3) DECIDES+. Participants in 'Usual Care' will continue to have access to their oncology health care team for questions related to cancer and cancer treatment, as per usual standard of care. Participants in both 'DECIDES' and 'DECIDES+' groups will receive access to DECIDES, and those in 'DECIDES+' will receive additional live, coach-assisted support. After 8 weeks, AYA and caregivers will complete a follow-up questionnaire and those in the 'DECIDES' and 'DECIDES+' groups will complete a semi-structured qualitative interview. Oncology clinicians of participating AYA will be invited to participate in a semi-structured qualitative interview. Researchers will compare groups to see if AYA and caregivers that receive access to DECIDES (with an informational handout vs. coach-assisted support) report more positive decision-making processes compared to those that receive standard of care.

DETAILED DESCRIPTION:
DECIDES is a developmentally appropriate, engaging, and interactive web-based decision support application that has been designed to address health literacy and includes:

* Education on cancer and cancer treatments, including clinical trials
* An exercise to identify perceived barriers and benefits to treatment options
* An exercise to clarify personal goals for treatment that align with life goals
* Resources to support communication with the oncology health care team

ELIGIBILITY:
Adolescent and Young Adults (AYA)

1. INCLUSION CRITERIA:

   * Ages 15-24 years old
   * Newly diagnosed or relapsed with leukemia/lymphoma, solid tumor, or brain tumor within 6 weeks of enrollment
   * Ability to read and speak English
   * If <18 Years Old: Parental/guardian permission to participate (informed consent)
2. EXCLUSION CRITERIA:

   * Inability to read or speak English
   * Pre-existing cognitive deficits (based on provider assessment) that result in impaired reading or decision-making capacity
   * AYA is a ward of the state or any other agency, institution, or entity
   * If <18 Years Old: No Parental/Guardian permission to participate (informed consent)

Caregivers

1. INCLUSION CRITERIA:

   * Parent or Legal Guardian of a participating AYA
   * Ability to read and speak English
2. EXCLUSION CRITERIA:

   * Foster parent or child advocate (i.e., caregiver is not biological parent or legal guardian)
   * Inability to read or speak English

Oncology Clinicians

1. INCLUSION CRITERIA:

   * Oncology clinician involved in decision-making about cancer treatment with enrolled AYA patients and caregiver(s)
   * Ability to read and speak English
2. EXCLUSION CRITERIA:

   * Oncology clinician that is not involved in decision-making about cancer treatment with enrolled AYA patients and caregiver(s)
   * Inability to read or speak English

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Barakat, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barakat LP, Hammer SN, Wen Y, Anil A, Schwartz LA, Reilly A, Bagatell R, Schapira MM, Li Y, Deatrick JA. Evaluation of a Decision Support Intervention for Adolescents and Young Adults Newly Diagnosed with Cancer: A Pilot Randomized Trial. MDM Policy Pract. 2025 Jun 26;10(1):23814683251344624. doi: 10.1177/23814683251344624. eCollection 2025 Jan-Jun. PMID 40584145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Potential participants were identified through outpatient oncology appointment and inpatient oncology unit lists at a single academic medical center between August 2020 and January 2023.
  * Adolescent and young adults (AYA) enrolled with a maximum of 2 caregivers, and those 18 or older could consent to participate independently.
  * Oncology clinicians were recruited to participate in an interview only; they were not randomized and did not complete assessments or provide demographics.
Pre-assignment Details: * n=117 (57 AYA, 47 Caregivers, 13 Oncology Clinicians) enrolled.
  * n=13 Oncology Clinicians were NOT randomized or administered a Baseline or Post-Intervention Assessment (per protocol).
  * n=7 (4 AYA, 3 Caregivers) were NOT randomized because they withdrew before randomization.
  * n=97 (53 AYA, 44 Caregivers) were randomized
Groups:
- Oncology Clinicians: Oncology Clinicians of participating AYA are not randomized to an intervention arm.
Period: Baseline
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Oncology Clinicians
Started (Total count of baseline assessments administered) | 21 | 35 | 41 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Started (AYA) (Count of baseline assessments administered to AYA) | 11 | 21 | 21 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Started (Caregivers) (Count of baseline assessments administered to Caregivers) | 10 | 14 | 20 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (AYA) (Count of baseline assessments completed by AYA) | 10 | 21 | 20 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (Caregivers) (Count of baseline assessments completed by Caregivers) | 10 | 14 | 20 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (Total count of baseline assessments completed) | 20 | 35 | 40 | 0 (Not Applicable (Baseline assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Period: Allocation to Group
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Oncology Clinicians
Started (Total count allocated to group.) | 21 (1 AYA had missing baseline data but was randomized with their enrolled caregiver.) | 35 | 41 (1 AYA had missing baseline data but was randomized with their enrolled caregiver.) | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Started (AYA) (Count of AYA allocated to group.) | 11 | 21 | 21 | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Started (Caregivers) (Count of Caregivers allocated to group.) | 10 | 14 | 20 | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Completed (AYA) (Count of AYA that completed participation in group.) | 11 | 20 | 20 | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Completed (Caregivers) (Count of Caregivers that completed participation in group.) | 10 | 14 | 19 | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Completed (Total count that completed participation in group) | 21 | 34 | 39 | 0 (Not Applicable (Oncology Clinicians are not allocated to a group).)
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Period: Post-Intervention Assessment
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Oncology Clinicians
Started (Total count of post-intervention assessments administered) | 21 | 34 | 39 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Started (AYA) (Count of post-intervention assessments administered to AYA) | 11 | 20 | 20 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Started (Caregiver) (Count of post-intervention assessments administered to caregivers) | 10 | 14 | 19 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (AYA) (Count of post-intervention assessments completed by AYA) | 10 | 18 | 20 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (Caregiver) (Count of post-intervention assessments completed by caregivers) | 9 | 13 | 19 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Completed (Total count of post-intervention assessments completed) | 19 | 31 | 39 | 0 (Not Applicable (Post-Intervention Assessments are completed by AYA and Caregivers and are not administered to Oncology Clinicians).)
Not Completed | 2 | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0
Period: Post-Intervention Qualitative Interview
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Oncology Clinicians
Started (Total count contacted to participate in qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 31 | 39 | 13 (Post-Intervention Assessments in PREVIOUS PERIOD are not administered to Oncology Clinicians.)
Started (AYA) (Count of AYA contacted to participate in qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 18 | 20 | 0
Started (Caregiver) (Count of Caregivers contacted to participate in qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 13 | 19 | 0
Completed (AYA) (Count of AYA that completed qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 15 | 18 | 0
Completed (Caregiver) (Count of Caregivers that completed qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 9 | 16 | 0
Completed (Total count of participants that completed qualitative interview) | 0 (Not Applicable. Participants in Usual Care did not receive the DECIDES intervention and do not participate in a Semi-Structured Qualitative Interview.) | 24 | 34 | 11
Not Completed | 0 | 7 | 5 | 2
Not completed — Lost to Follow-up | 0 | 7 | 5 | 0
Not completed — Started but did not finish due to time constraints. | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: * n=2 caregivers completed a Baseline Assessment but withdrew prior to randomization and are NOT reflected in the Overall Number of Baseline Participants count.
  * n=2 AYA had missing Baseline Assessment data but were randomized (1 Usual Care, 1 DECIDES+) with their caregiver, participated in the intervention, and completed the Post-Intervention Assessment; therefore, their demographic characteristics are included in the Overall Number of Baseline Participants count.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Total
Number analyzed (Participants) | 21 | 35 | 41 | 97
Age, Categorical [Count of Participants; unit: Participants] — Population: Two rows were added ('AYA' and 'Caregivers') to reflect the different type of participants in the overall population. AYA and Caregiver units were randomized together, to the same arm, but completed baseline and post-intervention measures separately (i.e., AYA-report and Caregiver-report).
  Participants
    AYA: number analyzed (Participants) | 11 | 21 | 21 | 53
    AYA: <=18 years | 7 | 13 | 13 | 33
    AYA: Between 18 and 65 years | 4 | 8 | 8 | 20
    AYA: >=65 years | 0 | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 10 | 14 | 20 | 44
    Caregivers: <=18 years | 0 | 0 | 0 | 0
    Caregivers: Between 18 and 65 years | 9 | 14 | 20 | 43
    Caregivers: >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two rows were added ('AYA' and 'Caregivers') to reflect the different type of participants in the overall population. AYA and Caregiver units were randomized together, to the same arm, but completed baseline and post-intervention measures separately (i.e., AYA-report and Caregiver-report).
  years
    AYA: number analyzed (Participants) | 11 | 21 | 21 | 53
    AYA | 17.3 (2.0) | 17.7 (1.4) | 17.5 (1.9) | 17.5 (1.7)
    Caregivers: number analyzed (Participants) | 10 | 14 | 20 | 44
    Caregivers | 47.0 (11.3) | 47.4 (6.0) | 49.7 (5.1) | 48.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two rows were added ('AYA' and 'Caregivers') to reflect the different type of participants in the overall population. AYA and Caregiver units were randomized together, to the same arm, but completed baseline and post-intervention measures separately (i.e., AYA-report and Caregiver-report).
  Participants
    AYA: number analyzed (Participants) | 11 | 21 | 21 | 53
    AYA: Female | 5 | 12 | 10 | 27
    AYA: Male | 6 | 9 | 11 | 26
    Caregivers: number analyzed (Participants) | 10 | 14 | 20 | 44
    Caregivers: Female | 10 | 11 | 15 | 36
    Caregivers: Male | 0 | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two rows were added ('AYA' and 'Caregivers') to reflect the different type of participants in the overall population. AYA and Caregiver units were randomized together, to the same arm, but completed baseline and post-intervention measures separately (i.e., AYA-report and Caregiver-report).
  Participants
    AYA: number analyzed (Participants) | 11 | 21 | 21 | 53
    AYA: Hispanic or Latino | 0 | 1 | 4 | 5
    AYA: Not Hispanic or Latino | 11 | 20 | 17 | 48
    AYA: Unknown or Not Reported | 0 | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 10 | 14 | 20 | 44
    Caregivers: Hispanic or Latino | 0 | 0 | 3 | 3
    Caregivers: Not Hispanic or Latino | 10 | 14 | 17 | 41
    Caregivers: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two rows were added ('AYA' and 'Caregivers') to reflect the different type of participants in the overall population. AYA and Caregiver units were randomized together, to the same arm, but completed baseline and post-intervention measures separately (i.e., AYA-report and Caregiver-report).
  Participants
    AYA: number analyzed (Participants) | 11 | 21 | 21 | 53
    AYA: American Indian or Alaska Native | 0 | 0 | 0 | 0
    AYA: Asian | 0 | 2 | 0 | 2
    AYA: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    AYA: Black or African American | 1 | 4 | 3 | 8
    AYA: White | 10 | 15 | 17 | 42
    AYA: More than one race | 0 | 0 | 1 | 1
    AYA: Unknown or Not Reported | 0 | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 10 | 14 | 20 | 44
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Caregivers: Asian | 0 | 1 | 0 | 1
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Caregivers: Black or African American | 1 | 1 | 3 | 5
    Caregivers: White | 9 | 12 | 15 | 36
    Caregivers: More than one race | 0 | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Decision Aid
Description: This is a 12-item study-team developed measure used to obtain acceptability ratings from AYA and caregivers (that completed participation in DECIDES or DECIDES+). This measure is based on The Ottawa Hospital's measure of acceptability regarding comprehension of components of a decision aid, its length, pace, amount of information, balance in presentation of information about options, and overall suitability for decision-making. Items are rated on a 5-point Likert scale (1=strongly disagree to 5=strongly agree). The average across 12 items is calculated to produce a total score that ranges from 1-5. Higher scores reflect greater acceptability. Two items related to the DECIDES Coach are not answered by participants in DECIDES who did not have access to a coach.
Time Frame: 8 weeks post-randomization
Population: NOTE. Measure was NOT administered to Usual Care group (per protocol).
  13 participants were excluded from analyses including:
  * n=8 non-protocol adherent participants (5 AYA, 3 Caregivers in the DECIDES group) that did not access the DECIDES intervention
  * n=1 Caregiver (in the DECIDES group) with missing data
  * n=2 non-protocol adherent participants (1 AYA, 1 Caregiver in the DECIDES+ group) that did not meet with the DECIDES Coach
  * n=2 Second Caregivers (in the DECIDES+ group)
Measure: Mean (Full Range); unit: Average Score on a Scale
Arm/Group | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 22 | 35
Average Score on a Scale
  AYA: number analyzed (Participants) | 13 | 19
  AYA | 4.10 [1 to 5] | 4.06 [1 to 5]
  Caregivers: number analyzed (Participants) | 9 | 16
  Caregivers | 4.01 [1 to 5] | 4.13 [1 to 5]

2. Primary Outcome: Usability of Decision Aid
Description: This is a 10-item scale collected from AYA and caregivers (that completed participation in DECIDES or DECIDES + coach) and oncology health care providers to measure perceptions of DECIDES usability. Items are rated on a 5-point Likert scale (1=strongly disagree to 5=strongly agree) and summed to produce a total score that ranges from 0 to 100. Scores are normalized to produce a percentile ranking. A score >80.3 reflects letter grade "A" (adjective rating "excellent"); 68-80.3 reflects letter grade "B" (adjective rating "good"), 68 reflects letter grade "C" (adjective rating "OK"); 51-67 reflects letter grade "D" (adjective rating "poor"); and <51 reflects letter grade "F" (adjective rating "awful").
Time Frame: 8 weeks post-randomization
Population: NOTE. Measure was NOT administered to Usual Care group (per protocol). Measure was administered to Oncology Clinicians during Interview.
  14 participants were excluded from analyses including:
  * n=8 (5 AYA, 3 Caregivers in the DECIDES group) that did not access the DECIDES intervention
  * n=2 (1 AYA, 1 Caregiver in the DECIDES+ group) that did not meet with the DECIDES Coach
  * n=2 Second Caregivers (in the DECIDES+ group)
  * n=2 Oncology Clinicians with missing data
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- No Arm/Group: Oncology clinicians were not allocated to an intervention arm. They completed the Systems Usability Scale during a qualitative interview.
Arm/Group | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | No Arm/Group
Number analyzed (Participants) | 23 | 35 | 11
Score on a scale
  AYA: number analyzed (Participants) | 13 | 19 | 0
  AYA | 75.96 (15.66) | 78.82 (13.90) |
  Caregivers: number analyzed (Participants) | 10 | 16 | 0
  Caregivers | 79.72 (12.77) | 83.33 (11.28) |
  Oncology Clinicians: number analyzed (Participants) | 0 | 0 | 11
  Oncology Clinicians |  |  | 86.98 (7.73)

3. Secondary Outcome: Perceived Involvement in Shared Treatment Decision-Making Process
Description: The SDM-Q-9 is a valid and reliable 9-item patient-reported questionnaire collected from AYA to measure their perceived involvement in the process of shared treatment decision-making with their oncology clinician. The physician version of the SDM-Q-9 (SDM-Q-Doc) was adapted for use with caregivers in this study to measure AYA involvement in shared decision-making with their oncology clinician, from the caregiver's perspective. Total scores range from 0 to 100. Higher scores reflect greater degree to which AYA were involved in a shared treatment decision-making process.
Time Frame: 8 weeks post-randomization
Population: 12 participants were excluded from analyses including:
  * n=8 non-protocol adherent participants (5 AYA, 3 Caregivers in the DECIDES group) that did not access the DECIDES intervention
  * n=2 non-protocol adherent participants (1 AYA, 1 Caregiver in the DECIDES+ group) that did not meet with the DECIDES Coach
  * n=2 Second Caregivers (in the DECIDES+ group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 57.33 (29.20) | 69.91 (17.06) | 69.26 (21.80)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 69.63 (24.06) | 77.78 (15.07) | 73.06 (20.83)

4. Secondary Outcome: Perceptions of Physician Engagement in Decision-Making Process
Description: This is a 5-item scale that measures AYA and caregiver perceptions of the extent to which clinicians engaged in five key elements of the decision-making process (e.g., discuss the available options with you in a way you could understand?, encourage you to ask questions or express any concerns you had about the available options?, involve you as much as you wanted in the decision making process?). The overall physician style score ranges from 0-100. Higher scores reflect more optimal communication with physician.
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 73.00 (22.14) | 92.31 (14.23) | 82.78 (27.18)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 76.67 (32.79) | 96.00 (9.66) | 95.00 (10.95)

5. Secondary Outcome: Knowledge of Cancer Clinical Trials
Description: This is a 25-item true/false questionnaire used to assess participant understanding of clinical trials and informed consent processes. Items are scored based on % correct, with higher scores reflecting more knowledge.
Time Frame: 8-weeks post randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Percent Correct
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 87.60 (5.48) | 81.85 (10.91) | 80.47 (14.62)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 87.56 (5.46) | 88.00 (7.21) | 88.31 (10.39)

6. Secondary Outcome: Attitudes Toward Cancer Clinical Trials
Description: This is a 35-item measure of AYA and caregiver attitudes toward clinical trials. Continuous scores were calculated from PRPQ items reflecting 'Perceived Benefits' (with a higher score suggesting positive attitudes) and from PRPQ items reflecting 'Perceived Barriers' (with a higher score suggesting negative attitudes). A 'Decision Balance' score was computed by converting the 'Perceived Benefits' and 'Perceived Barriers' scores to Z-scores, and then subtracting the 'Perceived Barriers Z-scores' from the 'Perceived Benefits Z-scores'. A 'Decision Balance' Z-score of 0 represents the population mean; a positive valence (3) reflects more positive attitudes to clinical trials and negative valence (-3) reflects more negative attitudes.
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Z-Score
  AYA: Decision Balance: number analyzed (Participants) | 10 | 13 | 19
  AYA: Decision Balance | 0.20 (1.35) | -0.15 (1.49) | 0.05 (0.91)
  Caregivers: Decision Balance: number analyzed (Participants) | 9 | 10 | 16
  Caregivers: Decision Balance | 0.03 (1.69) | 0.05 (1.87) | 0.33 (1.31)

7. Secondary Outcome: Uncertainty in Cancer Treatment Decision-Making Process
Description: This is a valid and reliable 16-item scale collected from AYA and caregivers to measure uncertainty in making cancer treatment decisions, including factors that contribute to uncertainty about cancer treatment options and perceptions of effective decision-making. Total scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 25.63 (12.68) | 23.44 (16.08) | 24.18 (20.36)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 25.00 (19.53) | 13.13 (12.93) | 20.02 (15.06)

8. Secondary Outcome: Regret About Cancer Treatment Decision-Making Process
Description: This is a valid and reliable 5-item scale collected from AYA and caregivers to measure distress or remorse about a cancer treatment decision. Total scores range from 0 (no regret) to 100 (high regret).
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 40.50 (32.87) | 27.31 (28.62) | 23.95 (24.24)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 17.78 (18.22) | 28.00 (35.76) | 13.13 (24.14)

9. Secondary Outcome: Satisfaction With Cancer Treatment Decision-Making Process
Description: This is a valid and reliable 6-item scale collected from AYA and caregivers to measure satisfaction with the cancer treatment decision that was made. Total scores range from 6 to 30, with higher scores reflecting higher satisfaction.
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 24.20 (3.49) | 25.23 (4.36) | 25.53 (4.45)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 24.89 (3.41) | 27.30 (3.23) | 26.44 (2.97)

10. Secondary Outcome: Self-confidence in Cancer Treatment Decision-Making Abilities
Description: This is a valid and reliable 11-item scale collected from AYA and caregivers to measure self-confidence in decision-making abilities. Total scores range from 0 (not confident) to 100 (extremely confident).
Time Frame: 8 weeks post-randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+)
Number analyzed (Participants) | 19 | 23 | 35
Score on a scale
  AYA: number analyzed (Participants) | 10 | 13 | 19
  AYA | 80.00 (14.60) | 78.15 (15.51) | 80.86 (16.02)
  Caregivers: number analyzed (Participants) | 9 | 10 | 16
  Caregivers | 81.06 (15.29) | 94.77 (8.09) | 86.93 (11.95)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Arm/Group | Usual Care | DECIDES With Informational Handout (DECIDES) | DECIDES With Coach-Assisted Support (DECIDES+) | Oncology Clinicians
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/35 | 0/41 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/35 | 0/41 | 0/13
Other Adverse Events (participants affected / at risk) | 0/21 | 0/35 | 0/41 | 0/13

LIMITATIONS AND CAVEATS:
Oncology Clinicians were not randomized to an intervention arm and did not participate in the intervention. Oncology Clinicians were enrolled to review DECIDES (live) during a semi-structured qualitative interview held via videoconference. Oncology Clinicians completed a measure of usability (Systems Usability Scale) during the interview. No other data were collected from Oncology Clinicians, including demographic data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT06191679/Prot_SAP_000.pdf